CLINICAL TRIAL: NCT05036356
Title: Burnout Reduction and Engagement App-based Trial of Headspace (BREATHE): A Randomized Clinical Trial
Brief Title: Burnout Reduction and Engagement App-based Trial of Headspace (BREATHE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Candace F. Granberg, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007153
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled App Group (Experimental): Subjects will receive access to the Headspace app and will receive weekly reminders to complete activities from the "Inspiration, Ideation, Implementation" block model of human-centered design in the app.
  Interventions: Other: Headspace App
- Ad lib App Group (Experimental): Subjects will receive access to the Headspace app and be encouraged to use it ad lib.
  Interventions: Other: Headspace App

INTERVENTIONS:
Other: Headspace App — A mobile-application ("app") focusing on teaching and sustaining mental well-being.

SUMMARY:
The purpose of this research is to develop a mobile app-based intervention to reduce burnout and improve well-being using human-centered design principles and stakeholder feedback.

DETAILED DESCRIPTION:
Recent studies of professional burnout among physicians have highlighted urology as a worrisome outlier: 39% of practicing urologists and 64% of urology residents reported high levels of depersonalization and emotional exhaustion. Despite the known association of burnout with adverse clinical outcomes, psychological distress, and career dissatisfaction, rigorous studies of physician-focused interventions remain limited.

Pilot studies of well-being mobile applications (e.g. headspace ®) have demonstrated better outcomes compared to traditionally delivered mindfulness interventions (e.g. in-person guided meditation). Nevertheless, a rigorous assessment of the impact of an app-based intervention on burnout is needed.

Therefore, the present study will assess the effectivity of a mobile app-based intervention to reduce burnout among healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Being a health-professional at the Urology Department of Mayo Clinic, RST
* Sign the informed consent and agreed to share data from the app to the research team.

Exclusion Criteria:

* Using an alternate app designed with the same purpose at the beginning, part and/or entire duration of the study.
* Not provide any data despite being included in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Change in burnout syndrome | Baseline, Week 12, Week 24
  Burnout levels among study population will be screened using the single-item burnout assessment tool for health care workers (West, Dyrbye, et.al. 2012) and the Professional Fulfillment Index (Trockel, et.al. 2018) . The single-item burnout tool has 2 questions with a 7-point Likert-type, frequency response scale (0 = never, 1 = a few times a year or less, 2 = once a month or less, 3 = a few times a month, 4 = once a week, 5 = a few times a week, 6 = every day) and cutoff values of 27 and 10 points, respectively. The Professional Fulfillment Index scales the answers of the items 7 to 16 from 0 to 4 (0 = not at all, 1 = very little, 2 = moderately, 3 = a lot, 4 = extremely) with a cutoff value of 1.33 points.
Change in professional fulfillment | Baseline, Week 12, Week 24
  Baseline professional fulfillment levels among study population will be screened using the 16-item Professional Fulfillment Index (Trockel, et.al. 2018) scaling the answers 1 to 6 from 0 to 4 (0 = not at all, 1 = somewhat true, 2 = moderately, 3 = very true, 4 = completely true) with a cutoff value of 3 points.

SECONDARY OUTCOMES:
User engagement metrics | Through study completion, approx. 24 weeks
  App-usage metrics will be characterized (user's platform usage), tracked continuously and compared between the intervention and control groups from baseline to follow-up phase (Week 24)
Qualitative knowledge and experience with app-based mindfulness practices | 24 Weeks
  Subject qualitative knowledge will measured by a self-reported questionnaire which asks participants to describe their previous experiences with well-being apps

CONTACTS AND LOCATIONS:
Overall Officials: Candace Granberg, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials